CLINICAL TRIAL: NCT03334344
Title: Using Virtual Reality (VR) Models for Preoperative Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceevra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20171006; NCT03421418 (obsolete NCT alias); NCT03534206 (obsolete NCT alias); NCT03542565 (obsolete NCT alias); NCT03556943 (obsolete NCT alias); NCT03666104 (obsolete NCT alias)
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2022-07

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Subjects whose surgeon will be viewing VR models in connection with the in addition to the source CT/MR image
  Interventions: Device: Ceevra Reveal
- Control Arm (No Intervention): Subjects whose surgeon will only be viewing CT/MR images in connection with the case

INTERVENTIONS:
Device: Ceevra Reveal — VR models generated using Ceevra Reveal are viewed by surgeons in connection with the case in addition to source CT/MR image.
  Arms: Intervention Arm

SUMMARY:
A prospective, randomized, controlled study designed to assess whether digital virtual reality (VR) models, created from existing CT scans and MRIs, provide surgeons with an improved understanding of their patients' anatomy, resulting in more efficient operations (robotic partial nephrectomy) and improved patient care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing robotic partial nephrectomy being performed by participating surgeon
* Subject is willing to be randomized between intervention and control arms

Exclusion Criteria:

* Cases involving subjects who are minors, pregnant or require an authorized representative for informed consent
* Cases in which the subject has a solitary or horseshoe kidney
* Cases in which the subject has more than two masses in the applicable kidney
* Cases involving a bilateral operation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russ Yoshinaka, BS, JD, Study Director — Sponsor GmbH
Locations (6):
- United States (6):
  - John Wayne Cancer Institute at Providence St. John's Heath Center, Santa Monica, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - University of Tennessee, Knoxville, Tennessee
  - Swedish Urology Group, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shirk JD, Thiel DD, Wallen EM, Linehan JM, White WM, Badani KK, Porter JR. Effect of 3-Dimensional Virtual Reality Models for Surgical Planning of Robotic-Assisted Partial Nephrectomy on Surgical Outcomes: A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911598. doi: 10.1001/jamanetworkopen.2019.11598. PMID 31532520

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 44 | 48
Completed | 44 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 44 | 48 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.7) | 57.6 (9.7) | 60.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 29 | 29 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 38 | 74
  Non-White | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 44 | 48 | 92

OUTCOME MEASURES:

1. Primary Outcome: Total Operative Time
Time Frame: During procedure
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
minutes | 163 [146.5 to 200] | 173.5 [148 to 199]

2. Secondary Outcome: Blood Loss
Time Frame: Measured at end of procedure
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
cc | 124.5 (90.5) | 145.7 (140.4)

3. Secondary Outcome: Clamp Time
Time Frame: Measured at end of procedure
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
minutes | 18 [12 to 22] | 18 [15 to 24]

4. Secondary Outcome: Number of Patients With Conversion to Open Surgery
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Participants | 0 | 0

5. Secondary Outcome: Number of Patients With Conversion to Radical Nephrectomy
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Participants | 3 | 3

6. Secondary Outcome: Number of Patients With an Intraoperative Complication
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Participants | 1 | 0

7. Secondary Outcome: Patient Hospital Stay
Time Frame: Measured at time of patient discharge, up to 10 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Days | 1.5 (0.8) | 1.64 (0.9)

8. Secondary Outcome: Number of Patients With a Positive Surgical Margin
Description: Incomplete removal of tumor as defined by the surgical pathology
Time Frame: Measured 1-2 weeks after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Participants | 0 | 0

9. Secondary Outcome: Post-Op Complication
Time Frame: Measured up to 6 months after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Participants | 4 | 2

10. Secondary Outcome: Readmission
Time Frame: Measured up to 6 months after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 44 | 48
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/48
Other Adverse Events (participants affected / at risk) | 0/44 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03334344/Prot_SAP_000.pdf